CLINICAL TRIAL: NCT04150328
Title: An Observational Retrospective Cohort Study of Lenalidomide Monotherapy in Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R/R DLBCL) to Generate a Historical Control for Clinical Trial MOR208C203 (RE-MIND)
Brief Title: Lenalidomide Monotherapy in R/R DLBCL
Acronym: RE-MIND
Status: Completed | Type: Observational
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Other Study IDs: MOR208C206
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study is designed to characterise the effectiveness of lenalidomide monotherapy in the treatment of R/R DLBCL and to compare the results with the efficacy outcomes of a tafasitamab-lenalidomide combination therapy in the clinical trial MOR208C203 (L-MIND)

DETAILED DESCRIPTION:
Tafasitamab (MOR00208) is currently in development for the treatment of R/R DLBCL. An ongoing, single-arm, phase II, open label, multicenter study (MOR208C203) is evaluating the efficacy and safety of tafasitamab combined with lenalidomide in patients with R/R DLBCL. In order to establish a lenalidomide monotherapy as a control cohort, this observational study aims to collect retrospective lenalidomide monotherapy data from real-world-evidence and to compare it with the tafasitamab-lenalidomide combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of DLBCL
* Relapsed/refractory to at least one previous systemic therapy for DLBCL
* Received at least one, but no more than three previous systemic regimens for the treatment of DLBCL, including at least one anti-CD20 containing therapy
* Received lenalidomide monotherapy for R/R DLBCL while being considered not eligible for an ASCT

Exclusion Criteria:

* CNS involvement by lymphoma
* Patients who received lenalidomide in combination with another anti-lymphoma therapy (including radiation)
* Previously treated with anti-CD19-targeted therapy or immunomodulatory drugs
* Patients who previously underwent allogeneic SCT
* Known simultaneous detection of MYC and BCL2 or BCL6 translocation according to FISH
* Patients with a history of other malignancies within 5 years prior to lenalidomide treatment start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: R/R DLBCL patients not eligible for HDC followed by ASCT who were treated with lenalidomide monotherapy
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Best overall/objective response rate (ORR) | Through study completion, an average of 9 months
  Proportion of patients with complete response (CR) or partial response (PR) as best response achieved at any time during the study

SECONDARY OUTCOMES:
Overall survival | Through study completion, an average of 9 months
  Time from treatment start until death from any cause
Complete response rate | Through study completion, an average of 9 months
  Proportion of patients having CR based on the best objective response achieved at any time during the study
Disease control rate | Through study completion, an average of 9 months
  Proportion of patients having CR, PR or stable disease (SD) based on the best objective response achieved at any time during the study

CONTACTS AND LOCATIONS:
Locations (49):
- United States (8):
  - MorphoSys Research Site, Rochester, Minnesota
  - MorphoSys Research Site, St Louis, Missouri
  - MorphoSys Research Site, Manhasset, New York
  - MorphoSys Research Site, New York, New York
  - MorphoSys Research Site, Rochester, New York
  - MorphoSys Research Site, Dublin, Ohio
  - MorphoSys Research Site, Charleston, South Carolina
  - MorphoSys Research Site, Greenville, South Carolina
- France (10):
  - MorphoSys Research Site, Bordeaux
  - MorphoSys Research Site, Le Mans
  - MorphoSys Research Site, Lille
  - MorphoSys Research Site, Lyon
  - MorphoSys Research Site, Paris
  - MorphoSys Research Site, Poitiers
  - MorphoSys Research Site, Pontoise
  - MorphoSys Research Site, Rouen
  - MorphoSys Research Site, Toulouse
  - MorphoSys Research Site, Tours
- Italy (28):
  - MorphoSys Research Site, Aviano
  - MorphoSys Research Site, Bergamo
  - MorphoSys Research Site, Bologna
  - MorphoSys Research Site, Brescia
  - MorphoSys Research Site, Como
  - MorphoSys Research Site, Cuneo
  - MorphoSys Research Site, Florence
  - MorphoSys Research Site, Meldola
  - MorphoSys Research Site, Milan
  - MorphoSys Research Site, Modena
  - MorphoSys Research Site, Napoli
  - MorphoSys Research State, Novara
  - MorphoSys Research Site, Padua
  - MorphoSys Research Site, Parma
  - MorphoSys Research Site, Pavia
  - MorphoSys Research Site, Perugia
  - MorphoSys Research Site, Piacenza
  - MorphoSys Research Site, Ponderano
  - MorphoSys Research Site, Ravenna
  - MorphoSys Research Site, Reggio Emilia
  - MorphoSys Research Site, Rimini
  - MorphoSys Research Site, Roma
  - MorphoSys Research Site, Salerno
  - MorphoSys Research Site, San Giovanni Rotondo
  - MorphoSys Research Site, Torino
  - MorphoSys Research Site, Udine
  - MorphoSys Research Site, Verona
  - MorphoSys Research Site, Vicenza
- Spain (3):
  - MorphoSys Research Site, Barcelona
  - MorphoSys Research Site, Madrid
  - MorphoSys Research Site, Salamanca